CLINICAL TRIAL: NCT03134079
Title: Influence on Food Liking of Adding Spices to Replace Dietary Sugar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: McCormick Science Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 14-1535
Record Dates: First submitted 2017-04-26; First posted 2017-04-28 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Taste Testing
Keywords: Taste Test; Spices; Reduced sugar; Food liking
MeSH Terms: interventions — Tea

STUDY DESIGN:
Intervention Model Description: Subjects were asked to taste test 3 versions of test items (in randomized order) and provide a liking score for each (tastings of each recipe were done on separate occasions separated by one week)
Who Masked: Participant
Masking Description: Subjects were blind to what version (recipe) of the taste test item they were tasting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- full sugar recipe (Active Comparator): Each subject was randomly assigned to one of six possible sequences to taste three recipes of each test item. Oatmeal and tea were served together and tastings occurred over three weeks; tasting of apple crisp occurred over three different weeks. Tastings of the three recipes occurred one week apart. The three recipes were full sugar recipe (FS), reduced sugar recipe (RS) and reduced sugar plus spice recipe (RSS). Each subject was randomly assigned to one of the below sequence schedules for each taste test whereby A, B, and C refer to one of the three recipes (FS, RS, or RSS):
  Sequence 1: A, B, C Sequence 2: A, C, B Sequence 3: B, A, C Sequence 4: B, C, A Sequence 5: C, A, B Sequence 6: C, B, A
  Interventions: Other: apple crisp; Other: tea; Other: oatmeal
- reduced sugar recipe (Experimental): Each subject was randomly assigned to one of six possible sequences to taste three recipes of each test item. Oatmeal and tea were served together and tastings occurred over three weeks; tasting of apple crisp occurred over three different weeks. Tastings of the three recipes occurred one week apart. The three recipes were full sugar recipe (FS), reduced sugar recipe (RS) and reduced sugar plus spice recipe (RSS). Each subject was randomly assigned to one of the below sequence schedules for each taste test whereby A, B, and C refer to one of the three recipes (FS, RS, or RSS):
  Sequence 1: A, B, C Sequence 2: A, C, B Sequence 3: B, A, C Sequence 4: B, C, A Sequence 5: C, A, B Sequence 6: C, B, A
  Interventions: Other: apple crisp; Other: tea; Other: oatmeal
- reduced sugar plus spice recipe (Experimental): Each subject was randomly assigned to one of six possible sequences to taste three recipes of each test item. Oatmeal and tea were served together and tastings occurred over three weeks; tasting of apple crisp occurred over three different weeks. Tastings of the three recipes occurred one week apart. The three recipes were full sugar recipe (FS), reduced sugar recipe (RS) and reduced sugar plus spice recipe (RSS). Each subject was randomly assigned to one of the below sequence schedules for each taste test whereby A, B, and C refer to one of the three recipes (FS, RS, or RSS):
  Sequence 1: A, B, C Sequence 2: A, C, B Sequence 3: B, A, C Sequence 4: B, C, A Sequence 5: C, A, B Sequence 6: C, B, A
  Interventions: Other: apple crisp; Other: tea; Other: oatmeal

INTERVENTIONS:
Other: apple crisp — Subjects tasted three items (apple crisp, tea and oatmeal) in a randomized sequence schedule to allow for tasting the three recipes (full sugar recipe, reduced sugar recipe and reduced sugar plus spice recipe) over three weeks. Oatmeal and tea were served together as a breakfast meal and tastings of oatmeal and tea were done over 3 weeks and tastings for apple crisp (served alone) were done over 3 different weeks. Subjects tasted one of the three recipes at each weekly seating.
Other: tea — Subjects tasted three items (apple crisp, tea and oatmeal) in a randomized sequence schedule to allow for tasting the three recipes (full sugar recipe, reduced sugar recipe and reduced sugar plus spice recipe) over three weeks. Oatmeal and tea were served together as a breakfast meal and tastings of oatmeal and tea were done over 3 weeks and tastings for apple crisp (served alone) were done over 3 different weeks. Subjects tasted one of the three recipes at each weekly seating.
Other: oatmeal — Subjects tasted three items (apple crisp, tea and oatmeal) in a randomized sequence schedule to allow for tasting the three recipes (full sugar recipe, reduced sugar recipe and reduced sugar plus spice recipe) over three weeks. Oatmeal and tea were served together as a breakfast meal and tastings of oatmeal and tea were done over 3 weeks and tastings for apple crisp (served alone) were done over 3 different weeks. Subjects tasted one of the three recipes at each weekly seating.

SUMMARY:
This study aims to reduce the amount of sugar in a particular food item and add spices to see if the food liking of that item rates as high or higher in a post meal survey. Through the weekly feeding and testing of the menu items the investigators will determine an opinion of the participants. Results of these surveys will determine whether participants enjoy the reduced sugar options as much as their full sugar counterparts.

DETAILED DESCRIPTION:
The Investigators will determine the overall consumer acceptability of a breakfast meal (tea and oatmeal) and a dessert (apple crisp) using a randomized, three-period, within subjects, crossover design. The three test conditions will be (1) Full sugar ("FS"), (2) reduced sugar (and calorie) with no added spice ("RS") and (3) reduced sugar (and calorie) plus spice ("RSS"). The two reduced sugar meals will be matched for calories. Subjects will taste each condition of the item on a separate day; tastings will be one week apart.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years

Exclusion Criteria:

* diagnosed taste or sensory disorders that would prevent subject from evaluating the food
* known eating disorders
* allergies to the test food/ingredients
* medical conditions that may adversely affect taste (e.g., dysgeusia)
* inability to complete the protocol
* personal dietary restrictions towards test meal items
* dislike of the particular food items to be served in the test meals
* Subjects who do not consume foods or beverages that contain sugar or to which they have added sugar will be excluded.
* Subjects who have not consumed or would not be willing to consume hot tea, oatmeal or baked apple products will be excluded.
* Subjects who are pregnant or trying to become pregnant will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2015-11-20 (Actual); Study Completion 2015-11-20 (Actual)

PRIMARY OUTCOMES:
9-point hedonic scale rating instrument to rate meal satisfaction | The day of tasting (once per week for 3 weeks)
  Overall liking of each meal with a 9-point hedonic scale rating instrument. The scale is a 9-point likert scale with scores ranging from 1 - 9 to assess liking (where the lowest rating of 1 indicated extreme disliking and the highest rating of 9 indicated extreme liking).

SECONDARY OUTCOMES:
9-point hedonic scale rating of the entree item (where applicable) | The day of tasting (once per week for 3 weeks)
  Overall liking of the entree item of each meal with a 9-point hedonic scale rating instrument for each item. The scale is a 9-point likert scale with scores ranging from 1 - 9 to assess liking (where the lowest rating of 1 indicated extreme disliking and the highest rating of 9 indicated extreme liking).
9-point hedonic scale rating of the beverage item (where applicable) | The day of tasting (once per week for 3 weeks)
  Over9-point hedonic scale ratingall liking of the beverage item of each meal with a instrument for each item. The scale is a 9-point likert scale with scores ranging from 1 - 9 to assess liking (where the lowest rating of 1 indicated extreme disliking and the highest rating of 9 indicated extreme liking).

CONTACTS AND LOCATIONS:
Overall Officials: John C. Peters, PhD, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krauss RM, Eckel RH, Howard B, Appel LJ, Daniels SR, Deckelbaum RJ, Erdman JW Jr, Kris-Etherton P, Goldberg IJ, Kotchen TA, Lichtenstein AH, Mitch WE, Mullis R, Robinson K, Wylie-Rosett J, St Jeor S, Suttie J, Tribble DL, Bazzarre TL. AHA Dietary Guidelines: revision 2000: A statement for healthcare professionals from the Nutrition Committee of the American Heart Association. Circulation. 2000 Oct 31;102(18):2284-99. doi: 10.1161/01.cir.102.18.2284. No abstract available. PMID 11056107
- [Background] Essed NH, Kleikers S, van Staveren WA, Kok FJ, de Graaf C. No effect on intake and liking of soup enhanced with mono-sodium glutamate and celery powder among elderly people with olfactory and/or gustatory loss. Int J Food Sci Nutr. 2009;60 Suppl 5:143-54. doi: 10.1080/09637480802710216. Epub 2009 May 21. PMID 19462326
- [Background] Howard BV, Wylie-Rosett J. Sugar and cardiovascular disease: A statement for healthcare professionals from the Committee on Nutrition of the Council on Nutrition, Physical Activity, and Metabolism of the American Heart Association. Circulation. 2002 Jul 23;106(4):523-7. doi: 10.1161/01.cir.0000019552.77778.04. No abstract available. PMID 12135957
- [Background] Trumbo P, Schlicker S, Yates AA, Poos M; Food and Nutrition Board of the Institute of Medicine, The National Academies. Dietary reference intakes for energy, carbohydrate, fiber, fat, fatty acids, cholesterol, protein and amino acids. J Am Diet Assoc. 2002 Nov;102(11):1621-30. doi: 10.1016/s0002-8223(02)90346-9. No abstract available. PMID 12449285
- [Background] Johnson RJ, Segal MS, Sautin Y, Nakagawa T, Feig DI, Kang DH, Gersch MS, Benner S, Sanchez-Lozada LG. Potential role of sugar (fructose) in the epidemic of hypertension, obesity and the metabolic syndrome, diabetes, kidney disease, and cardiovascular disease. Am J Clin Nutr. 2007 Oct;86(4):899-906. doi: 10.1093/ajcn/86.4.899. PMID 17921363
- [Background] King, SC, Snow, J, Meiselman, HL, Sainsbury, J, Carr, BT, McCafferty, D, Serrano, D, Gillette, M, Millard, L, Li, Q. Development of a questionnaire to measure consumer wellness associated with foods: The WellSense profile. Food Quality and Preference 39: 82-94, 2014.
- [Background] Littell, RC, Miliken, GA, Stroup, WW, Wolfinger, RD, Schabenberger, O, (eds.): SAS for Mixed Models, Second edn. Cary, NC: SAS Institute Inc, 2006.
- [Background] Malik VS, Popkin BM, Bray GA, Despres JP, Hu FB. Sugar-sweetened beverages, obesity, type 2 diabetes mellitus, and cardiovascular disease risk. Circulation. 2010 Mar 23;121(11):1356-64. doi: 10.1161/CIRCULATIONAHA.109.876185. No abstract available. PMID 20308626
- [Background] Peters JC, Polsky S, Stark R, Zhaoxing P, Hill JO. The influence of herbs and spices on overall liking of reduced fat food. Appetite. 2014 Aug;79:183-8. doi: 10.1016/j.appet.2014.04.019. Epub 2014 Apr 24. PMID 24769295
- [Background] Polsky S, Beck J, Stark RA, Pan Z, Hill JO, Peters JC. The influence of herbs, spices, and regular sausage and chicken consumption on liking of reduced fat breakfast and lunch items. J Food Sci. 2014 Oct;79(10):S2117-26. doi: 10.1111/1750-3841.12643. Epub 2014 Sep 12. PMID 25219391
- [Background] McGuire S. U.S. Department of Agriculture and U.S. Department of Health and Human Services, Dietary Guidelines for Americans, 2010. 7th Edition, Washington, DC: U.S. Government Printing Office, January 2011. Adv Nutr. 2011 May;2(3):293-4. doi: 10.3945/an.111.000430. Epub 2011 Apr 30. No abstract available. PMID 22332062
- [Result] Peters JC, Marker R, Pan Z, Breen JA, Hill JO. The Influence of Adding Spices to Reduced Sugar Foods on Overall Liking. J Food Sci. 2018 Mar;83(3):814-821. doi: 10.1111/1750-3841.14069. Epub 2018 Feb 24. PMID 29476623